2034-201-008

### STATISTICAL ANALYSIS PLAN

**Protocol Title:** A Phase 2b Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of AGN-151586 in Participants With Moderate to Severe Glabellar Lines

**Protocol Number: 2034-201-008** 

Compound Number: AGN-151586 (Botulinum Neurotoxin Serotype E, BoNT/E) for injection

**Short Title:** AGN-151586 Dose-Ranging Study for Treatment of Glabellar Lines

**Sponsor Name:** Allergan Sales LLC

Legal Registered Address: Allergan Sales LLC

5 Giralda Farms Madison, NJ 07940

**USA** 

Regulatory Agency Identifier Number(s): IND Number 130880

**Author:** 

**Version 1.0: 15 NOVEMBER 2019** 

Amendment 1: 13 OCTOBER 2020



| Table o | of Contents | 2 |
|---|---|---|
| List of | Tables | 3 |
| SAP V | Version History | 4 |
| 1. | Introduction | 5 |
| 1.1. | Objectives and Endpoints | 6 |
| 1.2. | Study Design | 10 |
| 2. | Statistical Hypotheses | 15 |
| 3. | Sample Size Determination | 16 |
| 4. | Populations for Analysis | 17 |
| 5. | Statistical Analyses | 18 |
| 5.1. | General Considerations | |
| 5.2. | Participant Disposition. | |
| 5.3. | Primary Effectiveness Endpoint Analysis | |
| 5.3.1. | Definition of Endpoint | |
| 5.3.2. | Main Analytical Approach | |
| 5.3.3. | Sensitivity Analysis | |
| 5.3.4. | Supplemental Approach. | |
| 5.4. | Secondary and Exploratory Effectiveness Endpoint Analyses | |
| 5.4.1. | Secondary and Exploratory Effectiveness Endpoints | |
| 5.4.2. | Main Analytical Approach | |
| 5.5. | Safety Analyses | 25 |
| 5.5.1. | Treatment Administration | 25 |
| 5.5.2. | Adverse Events | 25 |
| 5.5.3. | Clinical Laboratory Assessments. | 28 |
| 5.5.4. | Vital Signs | 29 |
| 5.5.5. | Electrocardiogram | 30 |
| 5.5.6. | Pregnancy Test Analyses | 30 |
| 5.6. | Other Analyses | 30 |
| 5.6.1. | Immunogenicity Analyses | 30 |
| 5.7. | Interim Analyses | 30 |
| 5.8. | Data Monitoring Committee (DMC) Analyses | 30 |
| 6. | Supporting Documentation | |
| 6.1. | Appendix 1 List of Abbreviations | |
| 6.2. | Appendix 2: Changes to Protocol-Planned Analyses | |
| 6.3. | Appendix 3: Supporting Study Information | |
| 6.3.1. | Demographics | |
| 6.3.2. | Baseline and Disease Characteristics | |
| 6.3.3. | Protocol Deviations | |
| 6.3.4. | Medical History | |
| 6.3.5. | Prior/Concomitant Medications | |
| 6.3.6. | Criteria for Potentially Clinically Significant Laboratory Results | 36 |

| 6.3.7.<br>6.4.1.<br>6.4.2.<br>6.4.2.1.<br>6.4.2.2.<br>7. | Criteria for Potentially Clinically Significant Vital Sign Results Data Handling Convention Analysis Window for Effectiveness and Safety Analyses Missing Date Imputation Missing/Incomplete AE Start Date Missing/Incomplete AE/Medication End Date References | |
|---|---|---|
| | List of Tables | |
| Table 1- | 1 Schedule of Activities | 12 |
| Table 4- | -1 Analysis Populations | 17 |
| Table 5- | 1 TEAE Tabular Summaries | 26 |
| | | 28 |
| Table 6- | 1 Protocol Deviation Summary | 35 |
| Table 6- | 2 Prior and Concomitant Medications | 36 |

## **SAP Version History**

This Statistical Analysis Plan (SAP) Amendment 1 for study 2034-201-008 is based on the Protocol Amendment 1 (dated 05 June 2020).

In addition to minor typographical corrections, other updates from the previous SAP version 1.0 (dated 15 November 2019) include the following:

- Section 1.1: Objectives and Endpoints table added based on objectives and endpoints stated in previous SAP. Estimand framework table updated
- Section 5.1: SAS version and MedDRA version updated to current versions. Added information about COVID-19-related reasons for modified visits to be reported as a listing.
- Section 5.3.2: Clarification provided for 95% confidence intervals that will be computed using the normal approximation (ie, Wald). In addition, p-values will be based on the stratified CMH tests, but the rate differences are not based on stratification.
- Section 5.5: Added that study period (prior to, during, after study intervention administration) will be presented for safety data listings.
- Section 5.5.2: Added a breakdown for treatment-related AEs to consist of study drug-related AEs and study procedure-related AEs. In addition, PDSOTs will be summarized as part of the overall AE table. Removed from summary the TESAEs leading to study discontinuation. Neurologic assessments will be summarized using descriptive statistics, and a listing will be provided. Treatment-emergent neurologic assessment-related AEs will also be presented by SOC and PT.
- Section 5.6.1: Updated immunogenicity analysis planned summary and stated that the results would be summarized if ready by time of the immunogenicity database lock.
- Sections 5.7 & 5.8: Stated that interim analyses are not applicable to the study, and the DMC analyses were moved to a separate section.
- Section 6.2: Added that a change to the protocol-specified analyses would be the summarization of TEAEs, not just AEs, per the primary safety endpoint.

2034-201-008

## 1. Introduction

This statistical analysis plan (SAP) provides a more technical and detailed elaboration of the statistical analyses of the efficacy and safety data as outlined and specified in study 2034-201-008 Protocol Amendment 1 (Approved version dated 05 June 2020). Specifications of tables, figures, and data listings are contained in a separate document.



# 1.1. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| Efficacy: To compare the efficacy between<br>placebo and a range of doses of AGN-151586<br>for the treatment of GL in participants with<br>moderate to severe GL | <ul> <li>Achievement of a ≥ 2-grade improvement<br/>from baseline on the FWS according to<br/>investigator assessments of GL severity at<br/>maximum frown at any postintervention<br/>timepoint through Day 7</li> </ul> |
| Safety: To compare the safety between<br>placebo and a range of doses of AGN-151586<br>for the treatment of GL in participants with<br>moderate to severe GL | Incidence of AEs; change from baseline in<br>hematology/chemistry/urinalysis laboratory,<br>vital sign, and ECG parameters; and presence<br>of antidrug antibodies |
| Secondary | |
| To compare the efficacy between placebo and<br>a range of doses of AGN-151586 for the<br>treatment of GL in participants with moderate<br>to severe GL, as measured by the FWS<br>(participant-assessed, investigator-assessed) | Achievement of a ≥ 2-grade improvement from baseline on the FWS according to participant assessments of GL severity at maximum frown at any postintervention timepoint through Day 7 |
| | <ul> <li>Achievement of a composite ≥2-grade<br/>improvement from baseline on the FWS at<br/>maximum frown as rated concurrently by the<br/>investigator and participant by timepoint</li> </ul> |
| | <ul> <li>Achievement of a ≥2-grade improvement from<br/>baseline on the FWS at maximum frown as<br/>rated by the investigator by timepoint</li> </ul> |
| | <ul> <li>Achievement of a ≥1-grade improvement from<br/>baseline on the FWS at maximum frown as<br/>rated by the investigator by timepoint</li> </ul> |
| | <ul> <li>Achievement of a ≥2-grade improvement from<br/>baseline on the FWS at maximum frown as<br/>rated by the participant by timepoint</li> </ul> |
| | <ul> <li>Achievement of a ≥1-grade improvement from<br/>baseline on the FWS at maximum frown as<br/>rated by the participant by timepoint</li> </ul> |
| | None or mild rating in FWS at maximum<br>frown as rated by investigator by timepoint |
| | None or mild rating in FWS at maximum<br>frown as rated by participant by timepoint |
| | Responders (defined by primary endpoint) achieving none or mild FWS at maximum frown as rated by the investigator by timepoint |





## **Estimand Framework:**

| Objective | | |
|---|---|---|
| Clinical | Statistical | |
| Category | Category | Estimand/Variable |
| Primary Objectiv | es: | |
| • Efficacy: | To compare the | efficacy between placebo and a range of doses of AGN-151586 for the |
| treatment of glabellar lines (GL) in participants with moderate to severe GL | | |
| Safety: To | o compare the saf | Fety between placebo and a range of doses of AGN-151586 for the treatment |
| of GL in | participants with | moderate to severe GL |
| Effectiveness <sup>1</sup> | Primary | <ul> <li>Variable: Achievement of a ≥ 2 grade improvement from baseline on<br/>the Facial Wrinkle Scale (FWS) With Photonumeric Guide according<br/>to investigator assessments of GL severity at maximum frown at any<br/>postintervention timepoint through Day 7</li> </ul> |
| | | <ul> <li>Population: The target population is the randomized population that has met the inclusion and exclusion criteria; the analysis population is the modified intention-to-treat (mITT) population (randomized participants who have received study intervention and have at least one postintervention measurement of investigator-rated FWS at maximum frown)</li> </ul> |
| | | <ul> <li>IES: Participants with no valid assessments at any postintervention timepoint through Day 7 will be excluded from the analysis</li> <li>PLS: Response rates between each dose group of AGN-151586 and</li> </ul> |
| _ | | <ul> <li>Analysis: Cochran-Mantel-Haenzsel (CMH) test stratified by baseline GL severity at maximum frown (investigator assessment), using observed data without imputation or adjustment for multiplicity.</li> <li>Between group comparisons will only be performed for each cohort's AGN-151586 group against the cohort's placebo group. Nominal pvalues will be presented for each statistical test.</li> </ul> |
| | Secondary | <ul> <li>Variables: Achievement of a none or mild grade on the FWS according to investigator assessment of GL severity at maximum frown at any postintervention timepoint through Day 7</li> <li>Population: The target population is the randomized population that has met the inclusion and exclusion criteria; the analysis population is the mITT population</li> <li>IES: Participants with no valid assessments at any postintervention timepoint through Day 7 will be excluded from the analyses</li> <li>PLS: Response rates between each cohort dose group of AGN-151586 and placebo</li> <li>Analysis: CMH test stratified by baseline GL severity at maximum frown using observed data without imputation or adjustment for multiplicity</li> </ul> |





IES = Intercurrent event(s) strategy; PLS = Population-level summary.

<sup>1</sup> All estimand attributes explicitly identified for primary/secondary and select key estimands only. Other secondary and exploratory estimands are similar.

## 1.2. Study Design

- This is a multicenter, double-blind, randomized, placebo-controlled, dose-escalation study to evaluate the safety and efficacy of a single study intervention cycle of AGN-151586 in participants with moderate to severe GL.
- Participants are adults 18 to 65 years old, with moderate to severe GL at maximum frown (as assessed by the investigator and participant using the FWS).
- Up to 5 doses of AGN-151586 will be evaluated and compared with placebo in a sequential cohort design, starting with the lowest dose.
- Each cohort will enroll a balanced distribution of participants with moderate or severe GL severity at maximum frown per investigator assessment (at least 40% and no more than 60% of either).
- The primary efficacy measure is the investigator's assessments of GL at maximum frown using the FWS.
- Participants will undergo a Screening Visit up to 30 days before randomization on Day 1. All screening data must be available to the investigator prior to randomization on Day 1.
- On Day 1, participants will be randomly assigned in a 3:1 ratio to receive AGN-151586 or placebo. Enrollment stratification will be by baseline GL severity at maximum frown, assessed by the clinician (principal investigator or physician subinvestigator) using the FWS.
- Study intervention on Day 1 will be administered as 5 injections in the glabellar complex (1 in the procerus and 2 in each corrugator).
- Participants will remain in the clinic for the first 12 hours after administration of study intervention for serial assessments at Hours 4, 8 and 12. Thereafter, participants return to the clinic on Day 2 (Hour 24 and Hour 36), Day 3 (Hour 48 and Hour 60), Day 7, Day 14, Day 21, Day 28, Day 35, and Day 42.
- For each dose group, an internal data monitoring committee (DMC), independent from the study team, will review select safety and efficacy data from a subset of participants (n ≥ 16) with data through 14 days postintervention (in addition to cumulative data from the prior cohort[s]).
- The DMC may recommend proceeding with the nominal dose for the next cohort, request additional data (eg, data from additional participants in the cohort, data from visits after Day 14), request to repeat the current dose or a lower dose, request an intermediate dose be evaluated (between the dose of the current cohort and the nominal dose for the next cohort), or request dose escalation be terminated.

2034-201-008



### The study scheme is as follows:



n = 40 per cohort at 3:1 randomization (AGN-151586:placebo)

The Schedule of Visits and Procedures during the study are presented in Table 1–1.



Table 1-1 Schedule of Activities

| Visit<br>Number | 1 | | 2 | | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | _ | | | | | 3 | - | | | ollow- | | , | 10 | 11 | End |
| Study Period | Screen ing (Days -30 to -1) | Randomiz<br>ation and<br>Study<br>Interventi<br>on<br>(Day 1) <sup>a</sup> | 1 | Day 1 | b | Do | y 2 | Do | у 3 | Da<br>y 7 | Da<br>y<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Da<br>y<br>35 | of<br>Study<br>(Day<br>42 or<br>Early<br>Exit) |
| Time after<br>administrati<br>on of study<br>intervention | | (Day 1) | 4<br>h | 8<br>h | 12<br>h | 24<br>h | 36<br>h | 48<br>h | 60<br>h | <b>y</b> 7 | 14 | 21 | 26 | 33 | |
| Visit<br>windows | | | ± 1<br>h | ±<br>1<br>h | ±<br>1 h | ± 2 h | ± 2 h | ± 2 h | ± 2 h | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>day |
| Consent/<br>authorization | X | | | | | | | | | | | | | | |
| Demographic s | X | | | | | | | | | | | | | | |
| Height and<br>weight | X | | | | | | | | | | | | | | |
| Inclusion/<br>exclusion<br>criteria | X | X | | | | | | | | | | | | | |
| Medical/surgi<br>cal history | X | | | | | | | | | | | | | | |
| | | X | | X | | X | | X | | X | X | X | X | X | X |
| | | X | | | | | | | | | | | | | |
| | | | | X | | X | | X | | X | X | X | X | X | X |
| | X | Х | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | х | Х | Х | X | X | X | X | Х | X | X | X | X | X | X |
| Standardized<br>facial<br>photography | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical examination <sup>d</sup> | X | X | X | | | X | | X | | X | X | X | X | X | X |



| Visit<br>Number | 1 | | 2 | | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Randomiz | | | | | | <u> </u> | Fo | ollow- | up | | <u> </u> | <u> </u> | End<br>of |
| Study Period | Screen ing (Days -30 to -1) | ation and Study Interventi on (Day 1) <sup>a</sup> | | <b>Day 1</b> | b | Da | y 2 | Da | y 3 | Da<br>y 7 | Da<br>y<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Da<br>y<br>35 | Study<br>(Day<br>42 or<br>Early<br>Exit) |
| Time after<br>administrati<br>on of study<br>intervention | | | 4<br>h | 8<br>h | 12<br>h | 24<br>h | 36<br>h | 48<br>h | 60<br>h | | | | | | |
| Visit<br>windows | | | ± 1<br>h | ±<br>1<br>h | ±<br>1 h | ± 2 h | ±<br>2 h | ± 2 h | ± 2 h | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>da<br>y | ± 1<br>day |
| Vital sign<br>measurement<br>s <sup>e</sup> | X | X | X | | | X | | X | | X | X | X | X | X | X |
| Neurologic assessments <sup>f</sup> | X | X | X | | | X | | X | | X | X | X | X | X | X |
| Urine pregnancy test (WOCBP) <sup>g</sup> | X | X | | | | | | | | | | | | | X |
| 12-lead ECGh | X | | | | | X | | X | | X | | | | | X |
| Collection of<br>blood and<br>urine samples<br>for<br>hematology,<br>chemistry,<br>and urinalysis<br>laboratory<br>testing <sup>i</sup> | X | | | | | | | X | | X | | | | | X |
| Collection of<br>blood<br>samples for<br>immunogenic<br>ity testing | X | | | | | | | | | X | | | X | | X |
| Adverse events | X | $\mathbf{X}^{\mathrm{j}}$ | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concurrent procedures | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |



| Visit<br>Number | 1 | | 2 | | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Randomiz | | | | | | | Fo | llow- | աթ | | | | End<br>of |
| | Screen<br>ing<br>(Days | ation and<br>Study<br>Interventi | | | | | | | | | Da | Da | Da | Da | Study<br>(Day<br>42 or |
| Study Period | -30 to<br>-1) | on<br>(Day 1) <sup>a</sup> | ] | Day 1 | b | Da | y 2 | Da | y 3 | Da<br>y 7 | у<br>14 | y<br>21 | y<br>28 | y<br>35 | Early<br>Exit) |
| Time after<br>administrati | | | | | | | | | | | | | | | |
| on of study<br>intervention | | | 4<br>h | 8<br>h | 12<br>h | 24<br>h | 36<br>h | 48<br>h | 60<br>h | | | | | | |
| Visit | | | | ± | | | | | | ±1 | ±1 | ± 1 | ±1 | ± 1 | |
| windows | | | ± 1<br>h | 1<br>h | ±<br>1 h | ± 2 h | ± 2 h | ±<br>2 h | ±<br>2 h | da<br>y | da<br>y | da<br>y | da<br>y | da<br>y | ± 1<br>day |
| Study<br>intervention<br>administratio<br>n | | X (0 h) | | | | | | | | | | | | | |

ECG = electrocardiogram;

GL = glabellar lines; WOCBP = women of childbearing potential

- All makeup must be removed and hair not obscuring the upper face prior to completing any assessment. All assessments must be completed before administration of study intervention at Hour 0.
- Participants must remain at the investigational site on Day 1 (ie, from baseline procedures through Hour 12 assessment).
- The investigator and participant must grade the severity of GL using the FWS at the same time, first at rest, then at maximum frown. The investigator and participant must not discuss their results with each other.
- A complete physical examination is to be done at the Screening Visit and EOS/Early Exit Visit. An abbreviated physical examination is be done at other visits. The abbreviated physical examination is limited to an examination of general appearance, heart, lungs, and abdomen.
- Vital sign measurements includes pulse rate, respiration rate, blood pressure, and body temperature. Participants are to be seated for at least 2 minutes before measurements are collected.
- The neurologic assessment includes the Focused Symptom Questionnaire and Focused Neurologic Examination.
- Women of childbearing potential (WOCBP) must have a negative pregnancy test at the Screening Visit and on Day 1 prior to randomization. The investigator may ask the participant to perform a urine pregnancy test at any time, which must be conducted at the investigational site. At each visit, site personnel must discuss with WOCBP and males with partners who are WOCBP compliance with contraceptive use.
- A 12-lead ECG will be taken with the participant in a semirecumbent position for ≥ 10 minutes before starting the tracing.
- Participant must be observed for at least 30 minutes after study intervention for adverse events.

## 2. Statistical Hypotheses

The following hypotheses will be used to compare each dose group of AGN-151586 with placebo within a cohort:

- Null hypothesis: AGN-151586 and placebo are equally effective in the probability of reducing GL severity at maximum frown as measured by a ≥ 2-grade improvement from baseline based on the investigator-rated FWS at any postintervention timepoint through Day 7.
- Alternative hypothesis: AGN-151586 and placebo are not equally effective in the probability
  of reducing GL severity at maximum frown as measured by a ≥ 2-grade improvement from
  baseline based on the investigator-rated FWS at any postintervention timepoint through
  Day 7.

The null and alternative hypotheses are as follows:

$$H_0$$
:  $P_{agn} = P_{pbo}$ 

$$H_a$$
:  $P_{agn} \neq P_{pbo}$ 

where  $P_{agn}$  and  $P_{pbo}$  are proportions of the participants with reduction in GL severity at maximum frown as measured by a  $\geq$  2-grade improvement from baseline based on the investigator-rated FWS at any postintervention timepoint through Day 7 for AGN-151586 group and placebo group, respectively.

The CMH test with stratification of baseline investigator-rated GL severity at maximum frown will be used to test the above hypothesis.



## 3. Sample Size Determination

The primary efficacy analysis will be conducted on the mITT Population, which consists of randomized participants who have received study intervention and have at least one postintervention measurement of investigator-rated FWS at maximum frown. A sample size of 40 participants per cohort will have approximately 88% power to detect a difference between an AGN-151586 dose group and the placebo group, assuming a 5% dropout rate and responder rates of 70% for the AGN-151586 study intervention group and 10% for the placebo group. The calculation is based on a 2-sided Chi-squared test (Fisher's exact test) with a 0.05 significance level using nQuery Advisor version 7.0.

For each cohort subset data reviewed by the DMC, beginning with the lowest dose before progressing to higher doses, the study will have increasing power to detect AE incidence among the participants treated with AGN-151586. For Cohort 1 DMC review, for example, with a subset of 12 participants treated with AGN-151586, there will be approximately 72% chance to detect an AE at a 10% incidence. For subsequent cohorts with increasing doses, for example, with subsets of 21 participants treated with AGN-151586, there will be approximately 90% chance to detect at AE at 10% incidence. A table is included below to show the range of probabilities of detecting AEs with varying incidence rates.

| TRUE | | | | |
|----------|--------------|--------------|--------------|--------------|
| EVENT | 12 on Active | 21 on Active | 30 on Active | 60 on Active |
| RATE (%) | Treatment | Treatment | Treatment | Treatment |
| 0.5% | 0.06 | 0.10 | 0.14 | 0.26 |
| | (0, 0.19) | (0, 0.23) | (0.02, 0.26) | (0.15, 0.37) |
| 1% | 0.11 | 0.19 | 0.26 | 0.45 |
| | (0, 0.29) | (0.02, 0.36) | (0.10, 0.42) | (0.33, 0.58) |
| 3% | 0.31 | 0.47 | 0.60 | 0.84 |
| | (0.05, 0.57) | (0.26, 0.69) | (0.42, 0.77) | (0.75, 0.93) |
| 5% | 0.46 | 0.66 | 0.79 | 0.95 |
| | (0.18, 0.74) | (0.46, 0.86) | (0.64, 0.93) | (0.90, 1) |
| 10% | 0.72 | 0.89 | 0.96 | >0.99 |
| | (0.46, 0.97) | (0.76, 1) | (0.89, 1) | (0.99, 1) |
| 20% | 0.93 | 0.99 | >0.99 | >0.99 |
| | (0.79, 1) | (0.95, 1) | (0.99, 1) | (0.99, 1) |
| 30% | 0.99 | >0.99 | >0.99 | >0.99 |
| | (0.92, 1) | (0.99, 1) | (0.99, 1) | (0.99, 1) |
| 50% | >0.99 | >0.99 | >0.99 | >0.99 |
| | (0.99, 1) | (0.99, 1) | (0.99, 1) | (0.99, 1) |



# 4. Populations for Analysis

The analysis populations will consist of participants as defined below:

Table 4–1 Analysis Populations

| Population | Definition | Study Intervention |
|---|---|---|
| mITT Population | All randomized participants who receive study intervention and who have at least one postintervention investigator-rated FWS measurement at maximum frown | As treated |
| Safety Population | All participants who receive study intervention | As treated |



#### **Statistical Analyses** 5.

#### 5.1. **General Considerations**

- The primary analyses will be performed after the database is locked and randomization schedule is released.
- The effectiveness endpoints will be analyzed based on the mITT Population. Safety analyses will be performed using the Safety Population. The analyses will be based on the actual study intervention that the participants receive.
- For each cohort, the effectiveness and safety endpoints will be analyzed/summarized by study intervention group, i.e., AGN-151586 group and placebo group, respectively. In addition, placebo groups across cohorts will be pooled to compare with each dose of AGN-151586 group as a sensitivity analysis.
- For applicable effectiveness and safety endpoints, baseline is defined as the last non-missing assessment prior to study intervention.
- Descriptive statistics for continuous variables include the sample size (N), mean, standard deviation, median, 1st and 3rd quartiles, minimum, and maximum. Summary statistics for categorical variables include the sample size (N), frequency count, and percentage.
- The primary analysis of the effectiveness endpoint, ie, the response rate of the participants with achievement of  $a \ge 2$  grade improvement from baseline on the FWS according to investigator assessments of GL severity at maximum frown at any postintervention timepoint through Day 7, will be analyzed using CMH tests stratified by baseline GL severity at maximum frown, to compare the between-group difference. The observed data without imputation will be used. Nominal p-values will be provided for each statistical testing. No multiplicity adjustment will be performed to control overall type I error.
- Summary of TEAEs, medical history, and concomitant medication will be summarized by study intervention group for each cohort. Also, the AGN-151586 groups across cohorts and the placebo groups across cohorts will be pooled.
- Partial dates will be treated as missing in computations, and will be listed in the data listings as they appear on the electronic case report form (eCRFs). No imputation of missing values will be performed, unless otherwise specified.
- The level of significance used for statistical testing of the effectiveness endpoints will be 0.05, 2-sided.



- The change from baseline values will be computed as the value for the postbaseline visit minus the baseline value.
- All statistical analysis will be performed using SAS version 9.4 or higher.
- Medical dictionary for regulatory activities (MedDRA) version 23.0 or higher will be used to code AEs and medical history.
- World Health Organization (WHO) Drug Dictionary will be used to code medications.
- Due to the COVID-19 pandemic, randomization into the study was curtailed for Cohort 3 only (38 of 40 participants randomized into Cohort 3), and visit assessments were modified for Cohorts 3 & 4 only. For Cohort 5, participants were expected to complete the visits as per the protocol; hence, no modifications were made to the visits for Cohort 5. These changes will be reported as a listing for modified visits due to COVID-19-related reasons.

#### 5.2. **Participant Disposition**

The number of participants in the study populations (mITT and Safety) will be summarized by study intervention group; the number of participants screened will be summarized overall.

Summary of study disposition will be provided by study intervention group for the following:

- Number of randomized participants
- Number of participants who receive study intervention
- Number of participants who discontinue the study
- Reasons for discontinuation of the study

#### 5.3. **Primary Effectiveness Endpoint Analysis**

#### 5.3.1. **Definition of Endpoint**

The assessments of the severity of GL at maximum frown using the validated FWS, is based on the following scale:

- 0 = None
- 1 = Mild
- 2 = Moderate
- 3 = Severe



investigator-rated FWS at maximum frown at any postintervention assessment through Day 7, he/she will be considered as a responder. The primary effectiveness endpoint is the response rate of the participants with achievement of a  $\geq$  2-grade improvement from baseline on the FWS according to investigator assessments of GL severity at maximum frown at any postintervention timepoint through Day 7.

#### 5.3.2. **Main Analytical Approach**

The proportion of responders for the primary endpoint will be analyzed based on mITT Population using CMH tests stratified by investigator assessment of baseline GL severity at maximum frown to compare each AGN-151586 study intervention group versus placebo for each cohort. In addition, placebo groups across cohorts will be pooled. Each AGN-151586 group will be compared against the pooled placebo groups as a sensitivity analysis. The observed data without imputation will be used.

The response rates of the participants with achievement of a  $\geq$  2-grade improvement from baseline on the FWS according to investigator assessments of GL severity at maximum frown at any postintervention timepoint through Day 7 will be calculated for each study intervention group. The corresponding 95% confidence intervals (CIs) using normal approximation (ie, Wald) will be provided.

The proportion difference, the corresponding Wald 95% CIs and nominal p-values will be provided for the comparison of response rates in the primary endpoint between different study intervention groups. P-values will be calculated based on the stratified CMH tests, but the rate differences are presented without stratification.

The p-values presented for each statistical test are deemed nominal. No multiplicity adjustment will be performed to control the overall Type I error.

#### 5.3.3. **Sensitivity Analysis**

Sensitivity analyses of the primary efficacy variable will be based on the non-responder imputation (NRI) method. If a participant does not have the valid investigator-rated FWS assessment at maximum frown at any postintervention assessment through Day 7, he/she will be considered as a non-responder. CMH tests stratified by baseline investigator assessment of GL severity at maximum frown will be used for the analysis based on the imputed data. In addition, the pooled placebo group will be compared to each AGN study intervention group for proportion differences for the primary analysis.

## 5.3.4. Supplemental Approach

Categorical descriptive statistics including the sample size (N), frequency count, and percentage for each response score and change from baseline will be provided by study intervention group and by visit. Change from baseline values will be computed as the value for the postbaseline visit minus the baseline value.

## 5.4. Secondary and Exploratory Effectiveness Endpoint Analyses

### 5.4.1. Secondary and Exploratory Effectiveness Endpoints

Secondary effectiveness endpoints include:

- Achievement of a ≥ 2-grade improvement from baseline on the FWS according to
   participant assessments of GL severity at maximum frown at any postintervention
   timepoint through Day 7
- Achievement of a composite ≥2-grade improvement from baseline on the FWS at maximum frown as rated **concurrently by the investigator and participant** by timepoint
- Achievement of a ≥2-grade improvement from baseline on the FWS at maximum frown as rated by the **investigator** by timepoint
- Achievement of a  $\geq$ 1-grade improvement from baseline on the FWS at maximum frown as rated by the **investigator** by timepoint
- Achievement of a ≥2-grade improvement from baseline on the FWS at maximum frown as rated by the **participant** by timepoint
- Achievement of a  $\geq$ 1-grade improvement from baseline on the FWS at maximum frown as rated by the **participant** by timepoint
- None or mild rating in FWS at maximum frown as rated by **investigator** by timepoint
- None or mild rating in FWS at maximum frown as rated by **participant** by timepoint
- Responders (defined by primary endpoint) achieving none or mild FWS at maximum frown as rated by the **investigator** by timepoint

AGN-151586

Exploratory effectiveness endpoints include:



CONFIDENTIAL AGN-151586 Statistical Analysis Plan Amendment 1 2034-201-008







### 5.4.2. Main Analytical Approach

The responder analyses will be analyzed in a similar way as for the primary effectiveness endpoint. The nominal p-values based on secondary effectiveness endpoints will be considered as supportive.

Descriptive statistics including the sample size (N), mean, standard deviation, median, 1st and 3rd quartiles, minimum, and maximum will be summarized by study intervention group and timepoint using the mITT Population for the FLO-11 item scores and total score, FLSQ item scores and domain scores.

### 5.5. Safety Analyses

Safety endpoints will be summarized by AGN-151586 dose group and placebo group in each cohort, as well as by total cohort groups and pooled placebo group and pooled AGN group using the Safety Population.

Study period in which events are experienced will be presented for safety data listings:

- 1 = screening period (prior to study intervention administration)
- 2 = treatment period (at time of study intervention administration)
- 3 = safety follow-up period (post-intervention through the end of study)

### 5.5.1. Treatment Administration

The treatment administration-related variables including the total dose will summarized by study intervention group using descriptive statistics.

Descriptive statistics will include the sample size (N), frequency count, and percentage for categorical endpoints, and sample size (N), mean, standard deviation, median, 1st and 3rd quartiles, minimum, and maximum for continuous endpoints.

### **5.5.2.** Adverse Events

An adverse event (AE) will be considered a treatment-emergent adverse event (TEAE) if:

- The AE began on or after the date and time of the study intervention; or
- The AE was present before the date and time of the study intervention, but increased in severity or became serious on or after the date and time of the study intervention.

A TEAE will be considered a treatment-emergent serious adverse event (TESAE) if it is a TEAE that is also a serious adverse event (SAE).

A TEAE will be considered a treatment-related TEAE if it is considered related to the study intervention or study procedures by the principal investigator.

The number and percentage of participants with TEAEs as well as the events in the following AE categories will be summarized by study intervention group, as well as for all participants who received AGN-151586, as described in Table 5-1.

If more than 1 AE is coded to the same preferred term for the same participant, the participant will be counted only once for that preferred term using the most severe and most related occurrence for the summarizations by severity and by relationship to study intervention.

Listings of all TEAEs, TESAEs, TEAEs leading to study discontinuation by participant, and death will be presented.

**Table 5-1 TEAE Tabular Summaries** 

| Endpoint | Description | Methodology |
|---|---|---|
| Overall summary | <ul> <li>Overall summary for the following categories:</li> <li>TEAEs</li> <li>Treatment-related TEAEs (including study drug-related TEAEs, study procedure-related TEAEs)</li> <li>TESAEs</li> <li>Treatment-related TESAEs</li> <li>Possible distant spread of toxin (PDSOT) TEAEs</li> <li>TEAEs leading to discontinuation from study</li> <li>Deaths</li> </ul> | Categorical descriptive summary statistics |
| TEAEs | <ul> <li>Overall summary and by system organ class (SOC) and preferred term (PT)</li> <li>Overall summary and by SOC, PT, and maximum severity</li> <li>Overall summary and by PT in descending order</li> </ul> | Categorical descriptive summary statistics |
| Treatment-related TEAEs • Study drug-related TEAEs • Study procedure- related TEAEs | <ul> <li>Overall summary and by SOC and PT</li> <li>Overall summary and by SOC, PT, and maximum severity</li> <li>Overall summary by maximum severity, duration, time to onset, resolution, and treatment required</li> </ul> | Categorical descriptive summary statistics, event descriptives |
| TESAEs | Overall summary and by SOC and PT if 5 or more participants overall reported such events | Categorical descriptive summary statistics |
| TEAEs leading to study discontinuation | Overall summary and by SOC and PT if 5 or more participants overall reported such events | Categorical descriptive summary statistics |

In addition, neurologic assessments (Focused Symptoms Questionnaire and Focused Neurologic Examination) will be reported using descriptive statistics for baseline, follow-up visits, and for



CONFIDENTIAL AGN-151586 2034-201-008

the entire study period. Listings will also be provided. Treatment-emergent neurologic assessment-related AEs will be identified based on the abnormal findings and reported by SOC and PT.

To assess possible distant spread of toxin (PDSOT), MedDRA preferred terms that may be associated with botulinum toxin effects have been identified. The number and percentage of participants reporting TEAEs that are included in the PDSOT term list will be tabulated. Summary tables will be provided for participants with TESAEs and participants with TEAEs leading to discontinuation if 5 or more participants reported such events. In addition, all PDSOT AEs will be listed by subject. The terms are listed below.



#### 5.5.3. **Clinical Laboratory Assessments**

Descriptive statistics for clinical laboratory values (in International System of Units [SI] units) and changes from the baseline values at each assessment visit will be presented by study intervention group for the following laboratory parameters:

Hematology: Absolute and differential white blood cell count (neutrophil count, lymphocyte count, monocyte count, basophil count, eosinophil count), hemoglobin, hematocrit, platelet count, red blood cell count, and red blood cell indices (mean corpuscular volume, mean



corpuscular hemoglobin, and mean corpuscular hemoglobin concentration, and distribution width).

Chemistry: Sodium, potassium, calcium, chloride, bicarbonate, magnesium, inorganic phosphate, glucose, blood urea nitrogen, creatinine, total protein, alkaline phosphatase (ALP), albumin, total bilirubin (TBL), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total cholesterol, yglutamyl- transferase (GGT), lactate dehydrogenase (LDH), Uric acid

Appearance, color, pH, specific gravity, glucose, protein, ketone, blood, urine Urinalysis: microscopy

Clinical laboratory test values will be considered potentially clinically significant (PCS) if they meet either the lower-limit or higher-limit PCS criteria listed in Table 6-3. The number and percentage of participants who have PCS postbaseline clinical laboratory values will be tabulated by study intervention group. The percentages will be calculated relative to the number of participants with available non-PCS baseline values and at least 1 postbaseline assessment. The numerator will be the total number of participants with available non-PCS baseline values and at least 1 PCS postbaseline value. A supportive tabular display of participants with PCS postbaseline values will be provided, including the PID number, baseline and all postbaseline (including non-PCS) values. In this listing, any participant with PCS value (if any) will also be included.

In addition, a tabular display showing all AEs that occurred in participants who had PCS postbaseline clinical laboratory values will be provided.

#### 5.5.4. **Vital Signs**

Descriptive statistics for vital signs (ie, temperature, respiratory rate, pulse rate, systolic and diastolic blood pressure) and changes from baseline values at each assessment visit will be presented by study intervention group.

Vital sign values will be considered as PCS if they meet both the observed-value criteria and the change-from-baseline criteria listed in Table 6-4. The number and percentage of participants with PCS postbaseline values will be tabulated by study intervention group. The percentages will be calculated relative to the number of participants with available non-PCS baseline values and at least 1 postbaseline assessment. The numerator will be the total number of participants with available non-PCS baseline values and at least 1 PCS postbaseline value. A supportive tabular display of participants with PCS postbaseline values will be provided, including the PID number, baseline and all postbaseline (including non-PCS) values.



In addition, a listing showing all AEs that occurred in participants who had PCS postbaseline vital sign values will be provided.

#### 5.5.5. Electrocardiogram

Electrocardiogram (ECG) evaluations by investigators are captured in the eCRF and are classified into 3 categories: normal, abnormal, or not evaluable. These data will be summarized by study intervention group as change from baseline for each parameter, as well as the number and percent of participants in each category for PCS. Data listings which include ECG basic parameters and any ECG abnormalities will be produced.

#### 5.5.6. **Pregnancy Test Analyses**

Urine pregnancy tests will be performed at the study center at screening, randomization/study intervention, and End of Study (Day 42 or Early Exit). Participants with a positive result will be presented in a listing for the Safety Population.

#### **Other Analyses** 5.6.

#### 5.6.1. **Immunogenicity Analyses**

Immunogenicity results, manifested as the presence of binding antibodies (positive), and neutralizing antibodies (positive) after a validated assay becomes available, to AGN-151586, will be summarized in a table for baseline and postbaseline, if available by immunogenicity database lock. Immunogenicity findings (positive) will be tabulated with the number and percentage of participants at each visit separately for each AGN-151586 treatment group. Percentages will be based on the number of treated participants with interpretable antibody assays in each treatment group at the specified visit.

#### 5.7. **Interim Analyses**

Not applicable.

#### **Data Monitoring Committee (DMC) Analyses** 5.8.

An internal DMC, independent from the study team, has been instituted to provide oversight in this study. Starting with Cohort 1, the DMC will convene to review select safety and efficacy data after the first subset of participants in Cohort 1 have completed the Day 14 visit. Following this review, the DMC will determine whether the study will proceed to Cohort 2 of dose escalation. After Cohort 2 proceeds, a similar review process will occur to determine whether Cohort 3 will proceed. This pattern repeats prior to the start of each new cohort. At each DMC review, data through Day 14 from a subset of participants ( $n \ge 16$ ) for any given cohort will be

CONFIDENTIAL AGN-151586 2034-201-008

reviewed. Additionally, cumulative data from participants from the prior cohort(s) will also be included in the DMC review.

At each DMC review, the DMC may recommend proceeding with the nominal dose for the next cohort, request additional data (eg, data from additional participants in the cohort, data from visits after Day 14), request to repeat the current dose or a lower dose, request an intermediate dose be evaluated (between the dose of the current cohort and the nominal dose for the next cohort), or request dose escalation be terminated.

The dose-escalation design of this study allows for careful review of select safety and efficacy data by the DMC to perform risk/benefit analyses prior to escalation to the next higher dose. Details of the activities and composition of the DMC are further described in the DMC charter.



AGN-151586

### **Supporting Documentation** 6.

AGN-151586

CONFIDENTIAL

## **6.1.** Appendix 1 List of Abbreviations

AE adverse event

ATC Anatomical Therapeutic Chemical

CI confidence interval

CMH Cochran-Mantel-Haenszel

DMC data monitoring committee

ECG electrocardiogram

eCRF electronic case report form

FWS Facial Wrinkle Scale With Photonumeric Guide

IES Intercurrent event(s) strategy

MedDRA medical dictionary for regulatory activities

mITT modified intention-to-treat

PCS potentially clinically significant

PDSOT possible distant spread of toxin

PLS Population-level summary

SAE serious adverse event

SAP statistical analysis plan

SI L Système International d'Unités (International System of Units)

SOC system organ class

TEAE treatment-emergent adverse event

TESAE treatment-emergent serious adverse event

WHO World Health Organization



# **6.2.** Appendix 2: Changes to Protocol-Planned Analyses

There is one change to the protocol-planned analyses. For the primary safety endpoints, TEAEs will be summarized, not AEs.

## 6.3. Appendix 3: Supporting Study Information

### 6.3.1. Demographics

Demographic parameters (age [years]; sex; race; ethnicity) will be summarized descriptively by study intervention group for the mITT and Safety Populations. Age (years) will be calculated relative to informed consent date.

### **6.3.2.** Baseline and Disease Characteristics

Baseline characteristics including weight, height, body mass index, and disease characteristics including baseline investigators' and participants' assessments of the severity of GL at maximum frown and at rest using the validated FWS, baseline FLO-11 and FLSQ scores will be summarized descriptively by study intervention group for the mITT Population.

### **6.3.3.** Protocol Deviations

Protocol deviations will be defined in a separate document. Unique participants reporting significant protocol deviations will be summarized in total and by treatment group for the mITT Population as described in Table 6-1.

Listing of significant protocol deviations will be provided.

**Table 6-1** Protocol Deviation Summary

| Endpoint | Description | Methodology |
|---|---|---|
| Significant protocol deviations | Number (%) of participants with significant protocol deviation will be summarized. | Categorical descriptive summary statistics |

### 6.3.4. Medical History

Abnormalities in participants' medical, surgical, cosmetic and dental history, encompassing abnormalities, surgeries, and procedures reported as occurring before the Screening Visit, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 23.0 or newer. The number and percentage of participants with abnormalities in medical and surgical histories in each system organ class and preferred term will be summarized by study intervention group for the mITT Population.

Listings will be provided for the mITT population.

### 6.3.5. Prior/Concomitant Medications

Medications will be coded using the WHO Drug Dictionary, version March 2017 or newer. Unique participants who reported medications (Anatomical Therapeutic Chemical [ATC] 4 class



and PT) will be summarized by study intervention group and by study period using the mITT Population as described in Table 6-2.

**Table 6-2** Prior and Concomitant Medications

| Endpoint | Description | Methodology |
|---|---|---|
| Prior medications | Medications taken before the date and time of study intervention | Categorical descriptive summary statistics |
| Concomitant medications | Medications on or after the date and time of study intervention to End-of-Study Visit (Day 42) | Categorical descriptive summary statistics |

## 6.3.6. Criteria for Potentially Clinically Significant Laboratory Results

Criteria for potentially clinically significant laboratory results are listing in Table 6-3.



Table 6-3 Criteria for Potentially Clinically Significant Laboratory Results

| Parameter | SI Unit | Lower Limit | Higher Limit |
|---|---|---|---|
| CHEMISTRY | • | • | |
| Albumin | g/L | < 0.9 × LLN | > 1.1 × ULN |
| Alanine aminotransferase (ALT) | U/L | _ | ≥ 3 × ULN |
| Alkaline phosphatase | U/L | _ | ≥ 3 × ULN |
| Aspartate aminotransferase (AST) | U/L | _ | ≥ 3 × ULN |
| Bilirubin, total | μmol/L | _ | > 1.5 × ULN |
| Calcium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Chloride | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Cholesterol, Total | mmol/L | | > 1.6× ULN |
| Creatinine | μmol/L | _ | > 1.3 × ULN |
| Glucose, fasting, serum | mmol/L | < 0.8 × LLN | > 1.4 × ULN |
| Glucose, random, serum | mmol/L | < 0.8 × LLN | > 1.4 × ULN |
| Potassium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Protein, total | g/L | < 0.9 × LLN | > 1.1 × ULN |
| Sodium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Urea Nitrogen (BUN) | mmol/L | _ | > 1.2 × ULN |
| HEMATOLOGY | | | |
| Basophils, absolute cell coun | t 10 <sup>9</sup> /L | | > 3 × ULN |
| Neutrophils, absolute cell count | 10 <sup>9</sup> /L | < 0.8 × LLN | > 1.5 × ULN |
| Hematocrit | Ratio | < 0.9 × LLN | > 1.1 × ULN |
| Hemoglobin | g/L | < 0.9 × LLN | > 1.1 × ULN |
| Platelet count | 10 <sup>9</sup> /L | < 0.5 × LLN | > 1.5 × ULN |
| Red blood cell count | $10^{12}/L$ | < 0.9 × LLN | > 1.1 × ULN |
| White blood cell count | 10 <sup>9</sup> /L | < 0.7 × LLN | > 1.5 × ULN |
| URINALYSIS | | | |
| pН | _ | < 0.9 × LLN | > 1.1 × ULN |
| Specific gravity | _ | _ | > 1.1 × ULN |

LLN = lower limit of normal value provided by the laboratory; SI = *Le Système International d'Unités* (International System of Units); ULN = upper limit of normal value provided by the laboratory.

## 6.3.7. Criteria for Potentially Clinically Significant Vital Sign Results

Criteria for potentially clinically significant vital sign results are listed in Table 6-4.



Table 6-4 Criteria for Potentially Clinically Significant Vital Sign Results

| Parameter | Flag | Criteria <sup>a</sup> | |
|---|---|---|---|
| | | Observed Value | Change From Baseline |
| Sitting systolic<br>blood pressure,<br>mm Hg | High | ≥ 160 | Increase of ≥ 20 |
| | Low | ≤ 90 | Decrease of ≥ 20 |
| Sitting diastolic<br>blood pressure,<br>mm Hg | High | ≥ 105 | Increase of ≥ 15 |
| | Low | ≤ 50 | Decrease of ≥ 15 |
| Sitting pulse rate,<br>bpm | High | ≥ 110 | Increase of ≥ 15 |
| | Low | ≤ 50 | Decrease of ≥ 15 |
| Weight, kg | High | _ | Increase of ≥ 7% |
| | Low | _ | Decrease of ≥ 7% |

a A postbaseline value is considered potentially clinically significant if it meets both the observed-value and the change-from-baseline criteria.

bpm = beats per minute.

# **6.4.** Data Handling Convention











#### 6.4.2.1. Missing/Incomplete AE Start Date

Imputation of dates with missing day and/or month is only applied to TEAEs. If adequate information is available, no imputation is needed. TEAE start dates with missing day or month will be imputed as following:

- If day and month are missing but year is the same as year of study intervention, then the imputed day and month will be the date of study intervention.
- If day is missing but the month and year are available, then the imputed day will be the first day of the month, or the date of study intervention, if they have the same month and year, whichever is later.

#### 6.4.2.2. Missing/Incomplete AE/Medication End Date

Imputation of dates with missing day and/or month is only applied to TEAEs when AE duration is calculated. If adequate information is available, no imputation is needed. TEAE end dates with missing day or month will be imputed as following:

• If day and month are missing but year is available, then the imputed day and month will be 31 Dec or the study exit date if they have the same year, whichever is earlier

If day is missing but the month and year are available, then the imputed day will be the last day of the month or the study exit date if they have the same month and year, whichever is earlier.

AGN-151586

#### 7. References

N/A